CLINICAL TRIAL: NCT06983145
Title: Study of the Postprandial Effect of Olive Leaf Biscuits and Tea Consumption on Plasma Antioxidant Status, as Well as on Metabolic Syndrome Indicators, in Healthy Individuals
Brief Title: Postprandial Effect of Olive Leaf Biscuits and Tea Consumption on Blood Biomarkers in Healthy Individuals
Acronym: OliherbCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Aegean (Other)
Responsible Party: Principal Investigator, ANTONIOS KOUTELIDAKIS, Associate Proffessor, University of the Aegean
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: OliherbCT
Record Dates: First submitted 2025-03-29; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Oxidative Stress; Inflammation Biomarkers
Keywords: olive leaf tea; olive leaf biscuits; inflammation; oxidative stress; acute clinical study
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Control: 2-3 pieces of biscuits with caramel coloring (total 120 g) and a glass (250 mL) of tea (natural mineral water with caramel coloring) for the control group Olive Leaf biscuit: 2-3 pieces of biscuits with 1.25 g. dried olive leaf powder (total 121.25 g) and a glass (250 mL) of tea (natural mineral water with caramel coloring) for the intervention group A and Olive leaf tea: 2-3 pieces of biscuits with caramel coloring (total 120 g) and a glass (250 mL) of tea (natural mineral water with 1.25 g. dried olive leaves) for the intervention group B.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): The individuals will consume 2-3 pieces of biscuits with caramel coloring (total 120 g) and a glass (250 mL) of tea (natural mineral water with caramel coloring) for the control group
  Interventions: Other: Olive Leaf tea
- Olive Leaf biscuit (Active Comparator): The individuals will consume 2-3 pieces of biscuits with 1.25 g. dried olive leaf powder (total 121.25 g) and a glass (250 mL) of tea (natural mineral water with caramel coloring)
  Interventions: Other: Olive Leaf tea
- Olive Leaf tea (Experimental): Individuals will consume 2-3 pieces of biscuits with caramel coloring (total 120 g) and a glass (250 mL) of tea (natural mineral water with 1.25 g. dried olive leaves)
  Interventions: Other: Olive Leaf tea

INTERVENTIONS:
Other: Olive Leaf tea — Individuals will consume 2-3 pieces of biscuits with caramel coloring (total 120 g) and a glass (250 mL) of tea (natural mineral water with 1.25 g. dried olive leaves)

SUMMARY:
This randomized controlled nutritional intervention study aims to investigate the bioactivity of dried olive leaves in biscuit and tea preparations, focusing on their postprandial effects on selected biomarkers and plasma antioxidant status. Healthy volunteers aged 18 to 65 from Limnos, Greece, will participate in the study, held at the Human Nutrition Unit of the University of the Aegean.

The study will last 15 days and features a cross-over design involving three groups:

Control Group: Consumes biscuits made with butter, flour, sugar, and caramel coloring, along with natural mineral water.

Intervention Group A: Receives the same biscuits with added dried olive leaf powder, accompanied by the same water.

Intervention Group B: Eats the standard biscuits with olive leaf tea instead of water. On each study day, participants will consume their meal over 15 minutes, followed by the liquid within 10 minutes. After a 7-day washout period, the groups will switch treatments for the second phase. The procedure will be repeated on the 15th day, ensuring that all participants experience each condition. Blood samples will be collected before and at 60, 120, and 240 minutes post-meal for analysis. Statistical processing will then be conducted to evaluate the effects on biomarkers and antioxidant status.

DETAILED DESCRIPTION:
This is the protocol of a randomized controlled nutritional intervention

- clinical study to investigate the bioactivity of preparations (biscuits and tea) with dried olive leaves. This is a nutritional intervention - clinical study of cross-over design (cross over design: acute study). The main objective of the study is to investigate the postprandial effect of olive leaves, on selected biomarkers and on the antioxidant status of plasma. The participants of the study will be healthy volunteers, aged 18-65 years, who will come from areas of Greece and will be based on the island of Limnos, in order to be able to be present on the days of the study. The study will be carried out in the specially designed space of the Human Nutrition Unit, University of the Aegean, in collaboration with external doctors. The total duration of the study will be 15 days (3 axes). Participants will be randomly divided into three groups. On the first day, the first group will consume a meal rich in carbohydrates and fats, which will consist of 2-3 biscuits made with butter, flour and sugar and drops of caramel coloring (E150a), along with a glass of natural mineral water with the addition of caramel coloring (E150a) at a refrigerator temperature of ~4°C (control group), the second group 2-3 biscuits made with butter, flour and sugar and dried olive leaf powder, along with a glass of natural mineral water with the addition of caramel coloring (E150a) at a refrigerator temperature of ~4°C (intervention group A) and the third group 2-3 biscuits made with butter, flour and sugar and drops of caramel coloring (E150a), along with a glass of tea made from dried olive leaves and natural mineral water at refrigerator temperature ~4°C (intervention group B). In all groups, the meal (control or intervention) will be consumed first and the liquid (control or intervention) will be consumed immediately afterwards. The total time for the meal (biscuits) will be 15 minutes and in the next 10 minutes, the liquid (olive leaf tea or water with caramel coloring) must also be consumed. After 7 days (washout period), the same volunteers will come to the specially designed area and the procedure will be repeated, with the difference that the control group on day 1 will belong to intervention group A, intervention group A will belong to intervention group B and intervention group B will belong to the control group. Finally, on the 15th day, the procedure will be repeated with the same volunteers, where the control group of the 1st day will now belong to the intervention group B, the intervention group A will belong to the control group and the intervention group B will belong to the intervention group A. On all 3 days, blood will be taken for analysis from the participants before, as well as 60, 120 and 240 minutes after the meals. Statistical processing of the results of the analyses will follow to present data regarding the postprandial levels of selected biomarkers and the antioxidant status of plasma.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, without underlying diseases (e.g. diabetes, cardiovascular, hypertension, hypercholesterolemia, hypertriglyceridemia, morbid obesity with BMI>40kg/m2)
* Aged 18-65 years at the start of the study
* Signed written consent to participate in the study and access by doctors to their medical history (diseases, medication)

Exclusion Criteria:

* People with a BMI >40
* Professional athletes
* People taking contraceptive treatment in the last 3 months
* People with a history of food allergy with hypersensitivity to any of the components of the administered product (e.g. milk protein or allergy-hypersensitivity to plants of the Oleaceae family) People taking supplements (e.g. antioxidants) or drugs that affect intestinal function (e.g. antibiotics) in the last 3 months or medication (hypoglycemic drugs or antihypertensive drugs or diuretics) that may interact with the administered product
* People taking any medication or supplement that may affect metabolism (e.g. GLP-1 analogues and receptor agonists, caffeine supplement, supplements weight loss/gain)
* Pregnant, lactating or menopausal women
* Individuals with substance abuse (drugs) or chronic alcoholism or total daily alcohol intake > 50 g/d
* Individuals with a chronic condition (history of cardiovascular disease, cancer, diabetes, hypertension, hyperlipidemia, neurological and neuropsychological disorders, active liver disease, severe renal dysfunction, severe stroke and conditions associated with increased risk of bleeding)
* Individuals with any other serious medical condition that may affect the individual's ability to participate in a nutritional intervention study.
* Individuals whose dietary preferences do not allow them to do so (e.g., vegetarians, vegans)
* Individuals who are not willing to comply with the study protocol and the periods of fasting and eating
* Individuals who are considered unreliable by the researcher or have a shorter life expectancy than the expected duration of the study, due to some disease or if they are in any condition that, in the opinion of the researcher, does not allow their safe participation in the study (drug addiction, alcohol abuse)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Total Antioxidant Capacity Concentration (mmol/L) | 1 hour, 2 hours, 4 hours
  Changes of Total Antioxidant Capacity Concentration from baseline
C- Reactive Protein Concentration (mg/dL) | 1 hour, 2 hours, 4 hours
  Changes of C-Reactive Protein Concentration from baseline

SECONDARY OUTCOMES:
Total Cholesterol Concentration (mg/dL) | 1 hour, 2 hours, 4 hours
  Changes of Total Cholesterol Concentration from baseline
High Density Cholesterol | 1 hour, 2 hours, 4 hours
  Changes of High Density Cholesterol from baseline
Low Density Cholesterol Concentration (mg/dL) | 1 hour, 2 hours, 4 hours
  Changes of Low Density Cholesterol Concentration from baseline
Glucose Concentration (mg/dL) | 1 hour, 2 hours, 4 hours
  Changes of Glucose Concentration from baseline
Triglycerides | 1 hour, 2 hours, 4 hours
  Changes of Triglycerides from baseline
Uric Acid Concentration (mg/dL) | 1 hour, 2 hours, 4 hours
  Changes of Uric Acid Concentration from baseline
Systolic Blood Pressure | 1 hour, 2 hours, 4 hours
  Changes of Systolic Blood Pressure from baseline
Diastolic Blood Pressure (mmHg) | 1 hour, 2 hours, 4 hours
  Changes of Diastolic Blood Pressure Concentration from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Lab of Human Nutrition and Public Health, Myrina, Limnos, Greece

IPD SHARING:
Plan to Share IPD: No
Due to sensitivity of data

DOCUMENTS (1):
  • Study Protocol (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT06983145/Prot_000.pdf